CLINICAL TRIAL: NCT01013961
Title: A Phase II Randomized Trial Comparing Standard and Low Dose Rituximab: Initial Treatment of Progressive Chronic Lymphocytic Leukemia in Elderly Patients Using Alemtuzumab and Rituximab
Brief Title: Rituximab and Alemtuzumab in Treating Older Patients With Progressive Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1908; E1908 (Other: ECOG-ACRIN Cancer Research Group); U10CA180794 (NIH)
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; small lymphocytic lymphoma; CLL; elderly; low dose rituximab; alemtuzumab; monoclonal antibodies
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (standard dose) (Active Comparator): Patients receive alemtuzumab subcutaneously (SC) on days 1-3, 6, 8, 10, 13, 15, 17, 20, 22, 24, 27, 29, and 31 and standard-dose rituximab 375 mg/m^2/week intravenously (IV) on days 8, 15, 22, and 29 in cycle 1 (33-day cycle). In cycle 2 and subsequent cycles (28-day cycle), patients receive alemtuzumab SC on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 and standard-dose rituximab IV on days 3, 10, 17, and 24. Treatment repeats every 28 days for up to 3 cycles.
  Alemtuzumab dose for cycle 1 week 1 requires a 'dose ramp' (3 mg day 1, 10 mg day2, and 30 mg day 3 of cycle 1) and then is 30 mg 3 times a week.
  Interventions: Biological: alemtuzumab; Biological: rituximab
- Arm B (low dose) (Experimental): Patients receive alemtuzumab SC on days 1-3, 6, 8, 10, 13, 15, 17, 20, 22, 24, 27, 29, and 31 and low-dose rituximab at 20 mg/m^2 IV on days 6, 8, 10, 13, 15, 17, 20, 22, 24, 27, 29, and 31 in cycle 1 (33-day cycle). In cycle 2 and subsequent cycles (28-day cycle), patients receive alemtuzumab SC and low-dose rituximab IV on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26. Treatment repeats every 28 days for up to 3 cycles.
  Alemtuzumab dose for cycle 1 week 1 requires a 'dose ramp' (3 mg day 1, 10 mg day2, and 30 mg day 3 of cycle 1) and then is 30 mg 3 times a week.
  Interventions: Biological: alemtuzumab; Biological: rituximab

INTERVENTIONS:
Biological: alemtuzumab — Given IV
Biological: rituximab — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab and alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer killing substances to them. Giving rituximab together with alemtuzumab may kill more cancer cells.

PURPOSE: This randomized phase II trial is studying two different doses of rituximab to compare how well they work when given together with alemtuzumab in treating older patients with progressive chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the rate of complete and overall response in elderly patients with progressive chronic lymphocytic leukemia (CLL) treated with one of two doses of rituximab combined with alemtuzumab to determine if the use of modified-dose rituximab significantly affects outcome.

Secondary

* To monitor and assess toxicity of these regimens.
* To determine the overall and progression-free survival, time to clinical response, time to next treatment, and duration of response in patients treated with these regimens
* To assess the correlation between risk stratification prognostic markers (i.e., CD38, ZAP-70, fluorescent in situ hybridization (FISH), and IgVH mutation) and clinical outcome.
* To assess response to these regimens using both the 1996 National Cancer Institute Working Group (NCI-WG 96) criteria and an expanded definition of response for patients in complete remission, including immunohistochemical examination of the bone marrow and sensitive flow cytometry (4-6 color) of blood for minimal residual disease and computed tomography (CT) scans for residual adenopathy.
* To determine the mechanism of action of rituximab and alemtuzumab and to determine mechanisms of resistance of a subpopulation of CLL cells to these drugs.

OUTLINE: This is a multicenter study. Patients are stratified according to FISH risk (low [13q14-] vs intermediate [12+, no abnormality, all other abnormalities] vs high [17p13-,11q22-]). Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive alemtuzumab subcutaneously (SC) on days 1-3, 6, 8, 10, 13, 15, 17, 20, 22, 24, 27, 29, and 31 and standard-dose rituximab intravenously (IV) on days 8, 15, 22, and 29 in cycle 1 (33-day cycle). In cycle 2 and subsequent cycles (28-day cycle), patients receive alemtuzumab SC on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 and standard-dose rituximab IV on days 3, 10, 17, and 24. Treatment repeats every 28 days for up to 3 cycles.
* Arm B: Patients receive alemtuzumab as in arm A. Patients also receive low-dose rituximab IV on days 6, 8, 10, 13, 15, 17, 20, 22, 24, 27, 29, and 31 in cycle 1 and on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 in cycless 2 and 3. Treatment repeats every 28 days for up to 3 cycles.

Blood and bone marrow samples are collected periodically for cytogenetic and biomarker analysis.

Alemtuzumab dose for Cycle 1 Week 1 of both Arms A and B requires a 'dose ramp' (3 mg day 1, 10 mg day2, and 30 mg day 3 of cycle 1).

After completion of study therapy, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL) meeting the following criteria:

  * Minimum threshold peripheral lymphocyte count of 5 x 10^9/L (CLL variant) OR palpable adenopathy > 1 cm or palpable splenomegaly 9small lymphocytic lymphoma [SLL] variant)
  * Immunophenotypic demonstrations of a population of B-lymphocytes (as defined by CD19+) that are monoclonal (by light-chain exclusion) AND have ≥ 3 of the following characteristics:

    * CD5+
    * CD23+
    * Dim surface light chain expression
    * Dim surface CD20 expression
  * FISH analysis is negative for immunoglobulin heavy chain/cyclin D1 gene (IGH/CCND1) and/or immunostaining is negative for cyclin D1 expression (to exclude mantle cell lymphoma)
* Progressive, symptomatic CLL, defined by at least one of the following:

  * Weight loss > 10% within the past 6 months attributable to progressive CLL (grade 2 or higher)
  * Extreme fatigue attributable to progressive CLL (grade 3 or higher)
  * Fevers > 100.5° F for 2 weeks without evidence of infection (grade 1 or higher)
  * Night sweats without evidence of infection (drenching)
  * Evidence of progressive bone marrow failure with hemoglobin < 11 g/dL or platelet count < 100 x 10^9/L
  * Rapidly progressive lymphadenopathy for which the largest node is ≤ 5 cm in any dimension

    * Largest lymph nodes involved in the neck, axilla, and groin need to be measured and followed for response

Exclusion Criteria:

* Prior treatment for CLL
* Massive splenomegaly > 6 cm below left costal margin, at rest, on clinical examination
* Lymphadenopathy > 5 cm in any diameter
* New York Heart Association class III or IV heart disease
* Recent myocardial infarction (within the past month)
* Uncontrolled infection
* Infection with the human immunodeficiency virus (HIV/AIDS)
* Serological evidence of active hepatitis B infection (HBsAg or HBeAg positive)
* Positive hepatitis C serology
* Evidence of active autoimmune hemolytic anemia, immune thrombocytopenia, or pure red blood cell aplasia
* Other active primary malignancy requiring treatment or that limits survival to ≤ 2 years, except for in situ carcinoma of the cervix or breast or non-metastatic basal cell or squamous cell carcinoma of the skin
* Major surgery within 4 weeks prior to pre-registration
* Concomitant use of continuous systemic corticosteroids

  * Prior corticosteroids are allowed but not at time of pre-registration to the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2015-04-14 (Actual); Study Completion 2015-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clive S. Zent, MD, Study Chair — University of Rochester
Locations (102):
- United States (102):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Mercy Clinic Cancer and Hematology - Rolla, Rolla, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Randolph Hospital, Asheboro, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - Danville Regional Medical Center, Danville, Virginia
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on October 8, 2010 and closed on October 31, 2013 with a total of 31 patients accrued. The first patient was accrued on April 27, 2011.
Pre-assignment Details: Peripheral blood (preferred) or bone marrow must be submitted at pre-registration for FISH risk analysis to determine stratification factor before randomization.
Period: Overall Study
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose)
Started | 16 | 15
Completed | 13 | 12
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose) | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Median (Full Range); unit: years] | 77 [67 to 92] | 76 [72 to 83] | 76 [67 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Complete Response (CR)
Description: Response was evaluated using NCI-WG96 criteria.
  A CR requires all of the following for >= 2 months:
  * Absence of lymphadenopathy > 1 cm in diameter by physical examination
  * No hepatomegaly or splenomegaly on physical exam
  * No constitutional symptoms
  * Normal complete blood count (CBC)
  * Patients achieving a clinical CR with negative CT scan after 2 cycles of therapy are re-evaluated using immunohistochemical examination of bone marrow biopsy for residual CLL cells. Patients with no evidence of residual disease and no radiological evidence of residual CLL on CT scan of chest-abdomen-pelvis and no clinical evidence of CLL on clinical evaluation after completion of 2 cycles of therapy will be considered to have a CR with no evidence of residual disease
Time Frame: Assessed after 2 cycles of treatment and 2 months after completion of therapy
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose)
Number analyzed (Participants) | 16 | 15
proportion of participants | 0.5 [0.247 to 0.753] | 0.4 [0.163 to 0.677]
Statistical Analysis 1: Comparison: Arm A (Standard Dose) vs Arm B (Low Dose); Test type: Superiority or Other; p = 0.722, Fisher Exact

2. Primary Outcome: Proportion of Patients With Overall Response (OR)
Description: OR is defined as either CR, clinical CR, or partial response (PR) evaluated by NCI-WG96 criteria. CR has been defined in the other primary endpoint.
  A clinical CR requires all of the following:
  * Absence of lymphadenopathy by physical examination
  * No hepatomegaly or splenomegaly. Spleen and/or liver, if considered enlarged at baseline, should not be palpable, due to disease, on physical exam
  * Absence of constitutional symptoms
  * Normal CBC as exhibited by:
  A PR requires all the following for ≥2 months:
  * ≥50% decrease in peripheral blood lymphocyte count from baseline
  * ≥50% reduction in lymphadenopathy
  * ≥50% reduction in size of liver and/or spleen
  * Polymorphonuclear leukocytes ≥1.5x10^9/L or 50% improvement over baseline
  * Platelets >100x10^9/L or 50% improvement over baseline
  * Hemoglobin >11.0 gm/dl or 50% improvement over baseline without transfusions
  * Any constitutional symptoms
Time Frame: Assessed after 2 cycles of treatment and 2 months after completion of therapy
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose)
Number analyzed (Participants) | 16 | 15
proportion of participants | 0.875 [0.617 to 0.985] | 0.933 [0.681 to 0.998]
Statistical Analysis 1: Comparison: Arm A (Standard Dose) vs Arm B (Low Dose); Test type: Superiority or Other; p = 1.0, Fisher Exact

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined to be time from randomization to death from any cause. Those still alive are censored at the date of last contact.
Time Frame: Assessed after 2 cycles of treatment, 2 months after completion of therapy and then yearly up to 5 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose)
Number analyzed (Participants) | 16 | 15
months | NA [22.3 to NA] — Median OS was not reached. The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [32.8 to NA] — Median OS was not reached. The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined to be time from randomization to progression (PD) or to death without documentation of progression. For patients without PD, follow-up is censored at the date of last disease assessment without PD, unless death occurs within three months following the date last known progression free.
  PD is characterized by at least one of the following:
  * ≥50% increase in the sum of the products of at least 2 lymph nodes on 2 consecutive examinations 2 weeks apart (at least 1 node must be >2 cm). Appearance of new palpable lymph nodes (>1 cm in diameter).
  * ≥50% increase in the size of liver and/or spleen as determined by measurement below the respective costal margin; appearance of palpable hepatomegaly or splenomegaly which was not previously present.
  * Absolute number of circulating lymphocytes with a count of >5x10^9/L
  * Transformation to a more aggressive histology
Time Frame: Assessed after 2 cycles of treatment, 2 months after completion of therapy and then yearly up to 5 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose)
Number analyzed (Participants) | 16 | 15
months | 12.8 [11.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 23.3 [14.8 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

5. Secondary Outcome: Time to Response
Description: Time to response is defined to be time from randomization to first confirmed CR, PR or clinical CR. Those without confirmed CR, PR or clinical CR are censored at the date of last disease assessment.
Time Frame: Assessed after 2 cycles of treatment, 2 months after completion of therapy and then yearly up to 5 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose)
Number analyzed (Participants) | 16 | 15
months | 4.8 [4.6 to 5.7] | 4.7 [2.7 to 6.5]

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined to be time from first confirmed CR, PR or clinical CR to progression or to death without documentation of progression. Patients without confirmed CR, PR or clinical CR are censored at time 0. Those without documentation of progression are censored at the date of last disease assessment without progression, unless death occurs within three months following the date last known progression free.
Time Frame: Assessed after 2 cycles of treatment, 2 months after completion of therapy and then yearly up to 5 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose)
Number analyzed (Participants) | 16 | 15
months | 9.8 [7.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 16.8 [10.1 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (Standard Dose) | Arm B (Low Dose)
Serious Adverse Events (participants affected / at risk) | 16/16 | 15/15
Other Adverse Events (participants affected / at risk) | 16/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Standard Dose) (N=16) | Arm B (Low Dose) (N=15)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Fatigue (General disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Serum sickness (Immune system disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 16 | 15
Lymphocyte count increased (Investigations) | 3 | 6
Neutrophil count decreased (Investigations) | 12 | 7
Platelet count decreased (Investigations) | 3 | 1
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 11 | 9
Investigations - Other, specify (Investigations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Nervous system disorders - Other (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Standard Dose) (N=16) | Arm B (Low Dose) (N=15)
Anemia (Blood and lymphatic system disorders) | 16 | 14
Atrial fibrillation (Cardiac disorders) | 0 | 1
Chills (General disorders) | 3 | 1
Fatigue (General disorders) | 8 | 7
Fever (General disorders) | 3 | 2
Injection site reaction (General disorders) | 2 | 1
Malaise (General disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Bladder infection (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 2 | 4
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 6 | 11
Lymphocyte count increased (Investigations) | 7 | 7
Neutrophil count decreased (Investigations) | 9 | 8
Platelet count decreased (Investigations) | 11 | 10
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 13 | 15
Anorexia (Metabolism and nutrition disorders) | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less